CLINICAL TRIAL: NCT03142984
Title: A Randomized Controlled Trial of Gentle Touch/Early Massage With a New Wash and Lotion Regimen for Improved Skin Barrier Strength, Parental Bonding, and Physical Development in Newborn Babies: The Barrier Optimizing Skincare for Newborn Development (BOND) Trial
Brief Title: UK Baby Study Using a Baby Wash and Lotion Regimen
Acronym: BOND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been on hold due to the COVID-19 pandemic. As of Mar 23, 2022, the Sponsor has decided to terminate the study for administrative reasons.
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CO-1610 1411 2628-SBCT; CO-161014112628-SBCT (Other: Johnson & Johnson)
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Newborns
MeSH Terms: interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): An open use test in a cohort of newborn babies to confirm the tolerability and evaluate the acceptability of a new Baby Wash & Shampoo product and Baby Lotion.
  Baby Wash & Shampoo (F# 13217-070) Baby Lotion (F# 13217-071)
  Interventions: Other: Cosmetic Products
- Phase 2 (Experimental): An evaluator blind, randomized, controlled trial to determine whether a wash and lotion regimen used for 12 weeks can strengthen the skin barrier in newborns when compared to standard skincare practices without massage.
  Baby Wash & Shampoo (F# 13217-070) Baby Lotion (F# 13217-071)
  Interventions: Other: Cosmetic Products

INTERVENTIONS:
Other: Cosmetic Products — Phase 1:
  Baby Wash & Shampoo (F# 13217-070) Baby Lotion (F# 13217-071)
  Phase 2:
  Baby Wash & Shampoo (F# 13217-070) Baby Lotion (F# 13217-071)

SUMMARY:
The skin of a newborn has a sensitive skin barrier relative to an older child and an adult. Newborn's skin, for example, is extremely vulnerable to damage by environmental agents such as harsh detergents, some topical oils, and other irritant chemicals. Evolving perspectives on barrier dysfunction in newborn babies has led to the idea that there may be a window of opportunity in the first few months of a newborn's life to change the environmental agents that their skin is exposed to in order to maximize skin health. These environmental changes could involve the use of optimally formulated wash products and emollients, as well as the removal of all other irritant substances that could damage the skin barrier. Further research is required to identify skincare practices that are harmful and those that are positive, and to ultimately ascertain what the optimum skincare routine should be.

An important skincare strategy is to identify an appropriate regimen (use of topical emollients and wash products) that will be used to maintain healthy skin in the future. Baby massage in particular has been shown to enhance the bond between mother and newborn, highlighting that early intervention can support skin health while also being a rewarding experience.

Gentle Touch/Early Massage:

Apply the lotion with a gentle touch to communicate love to your baby and to create a special bonding moment with skin-to-skin touch. Your touch nurtures baby's social, emotional and physical development. Please take your time to apply consciously the lotion on the whole body of your baby while engaging with her/him. Your touch, light but present, will be consistent across all the face and body areas, it is delicate and soft but more than just applying the lotion.

Parents/guardians are using products to help care for their newborn's skin and there is a need to help parents/guardians identify the most appropriate products through research. This study aims to help address this need.

DETAILED DESCRIPTION:
2 BACKGROUND 2.1 SKIN DEVELOPMENT FROM BIRTH The skin visually reaches maturity anywhere between 30 and 37 weeks of gestational age, yet neonatal and infant skin exhibits a 'sensitive' nature.1 To emphasize this, 78% of participants in one study reported a 'rash' in the first month of their newborns life.2 Its now clear that this sensitivity is related to the functioning of the skin barrier, formed by the skins uppermost layer, the stratum corneum. It takes more than 12 months following birth before the stratum corneum reaches structural maturity at a microscopic level.3 This is reflected by the reduced function of the skin barrier during this time, indicated by elevated transepidermal water loss (TEWL).4 The reduced skin barrier function exhibited during the months following birth increases the risk of irritant and allergen penetration through the skin and consequently the development of dermatological conditions.

2.2 SKIN CLEANSING For both children and adults, bathing to cleanse the skin is a hygienic necessity. The goal of hygiene is the preservation of skin health. Cleansing is essential to remove: potentially pathogenic bacteria, such as those from faeces; bodily secretions, such as faeces and saliva that contain enzymes (lipases and proteases) that breakdown the skin barrier; foods, including milk that can disturb skin homeostasis and peanuts that can cause sensitization; and other chemical irritants in the environment.1 However there is a balance to be made between cleansing the skin and preservation of its homeostatic properties such as skin barrier function and integrity.5 For instance some soaps and cleansers used to clean the skin that contain harsh detergents, such as sodium lauryl sulfate (SLS), increase skin surface pH, reduce skin hydration and alter skin barrier function.6 Nevertheless cleansers are important. Washing with water alone is ineffective at removing fat-soluble substances from skin.7 The surfactants in cleansers are required to remove these potential fat-soluble irritants. Moreover, washing with tap water alone leads to the extraction of water-soluble metabolites from the skin, including NMF, and causes mild irritation and increased skin dryness. Washing with hard water, as opposed to soft water, in particular is consistently reported to increase the risk of developing AD. A balance is therefore required between effective cleansing and the need for cleansers that are kind to the skin.8 There is now a wide range of detergents and detergent complexes available for the use in cleansing with a spectrum of effects on the skin from harsh irritant effects, such as those caused by SLS, to very mild effects comparable to washing with water alone.

The use of cleansing products compared to water alone for bathing babies has been subject to a systematic review,9 which focused on two trials. One study10 comprised of four trial arms, including washing twice weekly with a wash gel product; bathing twice weekly with water then applying a cream; bathing with wash gel and applying cream after bathing; and bathing with water only. The second study11 compared two different liquid cleansers with water for bathing infants. The results of these studies indicated no harm to skin barrier function with the tested cleaning agents, although the number of babies in each treatment arm was small.9 A large UK-based trial of a mild pH 5.5 liquid SLS-free cleanser versus water alone in bathing newborn babies for the first 28 days, conducted since this systematic review, showed essentially no differences in TEWL, hydration, skin surface pH and clinical observations.12 Skin hydration was raised in the cleanser arm at 14 days postnatal (ITT: mean wash score 49.7 (SD 9.2) vs. water 46.7 (SD 8.4), p=0.02, 95% CI -5.46 to -0.43), but was equal to those in the water group at 28 days postnatal. The evidence suggests that while some cleansers, particularly those containing SLS, can be harsh on the skin, other cleansers are available that have very mild effects on the skin, effects as least as mild as washing with water alone. The advantage of these mild cleansers is their increased cleansing efficacy and cosmetic acceptability. Given the limited number of robust clinical trials in this area there is a need to conduct further research to enable healthcare professionals and parents/carers to identify suitable and safe wash products and cleansing regimens for their babies and infants.

2.3 CURRENT GUIDANCE ON SKIN CLEANSING Current guidance on skin cleansing has been limited by the lack of available high quality evidence, leading to a number of differing guidelines.13-17 Hence, there has been confusion amongst health professionals in relation to appropriate advice.18 Guidance from the World Health Organization13 is limited to bathing a baby in warm water, at least 6 hours following birth. There is no United Kingdom NICE (National Institute for Clinical Excellence) guidance specifically about neonatal skin care. The NICE Postnatal Care Guidelines17 contains one paragraph about neonatal skin care which recommends that cleansing agents, lotions or medicated wipes should not be used; using only a mild non-perfumed soap where necessary. No evidence is cited to support this practice, and recent trials have demonstrated that the use of products can significantly reduce the development of dermatological conditions. In contrast to the NICE Postnatal Care Guideline, AWOHNN14,19 guidance is more comprehensive and specific and recommends use of a cleansing wash, with a neutral pH, that has been specifically formulated for use on babies.

Although there are guidelines available, not all are evidence based and debate still remains on best practice. The most recent guideline, produced by a panel of experts, advocates the use of wash products. Based upon this guideline the recently NHIR-funded Barrier Enhancement for Eczema Prevention (BEEP) study investigating an early skincare intervention in babies provided the following advice to participants: (1) avoid soap and bubble bath; (2) use a mild, fragrance-free synthetic cleanser designed specifically for babies; (3) avoid bath oils and additives; (4) use a mild, fragrance-free shampoo designed specifically for babies and avoid washing the suds over the baby's body; and (5) avoid using baby wipes, where possible.20 The challenge for parents is identifying 'mild' products, and so this advice currently has limited real-world value until more evidence on the effects of different products becomes available. There have been substantial advances in formulation technology of baby wash products since some of these guidelines were written highlighting the need for further research into neonatal skincare practices.10-12,21-24 2.4 INFANT SKIN MASSAGE Infant massage is a traditional practice advocated and used throughout the world to promote physical and mental development.25 Moreover it is an integral aspect of topical emollient use in newborn babies because emollient lotions and creams applied to the skin must be rubbed, or 'massaged', in. In the UK more than half of maternity/neonatal units endorse the use of massage oil as part of infant skincare.26 A number of studies into infant massage have identified potential physical and mental benefits that require validation.25 These benefits include: increased weight, length, head circumference; improved sleep; reduced episodes of crying/fussing; improved motor skills (gross and fine); enhanced personal and social behavior; and improved psychomotor development. The development of a secure attachment between parent and infant in the early years is highly protective in promoting healthy psychosocial and emotional development. Infant massage may have a role in facilitating the development of early sensitive parent - infant relationships and attunement, known precursors to the development of secure attachments27. At 2 months of age the hypothalamic-pituitary-adrenocortical system produces and regulates glucocorticoid cortisol in response to stress. Sensitive and attuned parents-infant interactions are associated with reduced cortisol excretion and thus improved affect regulation in infants28. A randomized controlled trial conducted by Gurol and Polat on infant massage in 120 newborn babies found a significant positive effect of the intervention on attachment between the mother and baby.29 The association between early secure attachment relationships, and the promotion of healthy brain development, emotional wellbeing and mental health is increasingly recognized and associated with improved outcomes for children across all domains of functioning30. Although there is significant research in the area of infant / child massage which supports positive benefits, very few studies have specifically studied the effects of massage in combination with a specific product form as a focus of the study.

Gentle Touch/Early Massage:

Apply the lotion with a gentle touch to communicate love to your baby and to create a special bonding moment with skin-to-skin touch. Your touch nurtures baby's social, emotional and physical development. Please take your time to apply consciously the lotion on the whole body of your baby while engaging with her/him. Your touch, light but present, will be consistent across all the face and body areas, it is delicate and soft but more than just applying the lotion.

Improved parent-infant interaction is currently an overlooked potential benefit of emollient use in newborn babies in most studies reported. Care is needed when selecting an emollient medium for infant massage because some topical oils have been found to damage the skin barrier.31-33 This study aims to investigate the effects of an emollient lotion specially formulated for use in newborns.

2.5 PATIENT AND PUBLIC INVOLVEMENT We have taken the views of parents with young babies into consideration when developing this study so that the findings have the greatest meaning and impact to them. In 2008 the views of 26 mothers, 20 midwives and 10 health visitors on baby bathing practices were ascertained as part of a qualitative study.18 Since then we have gathered the views of parents on baby bathing practices and clinical research on these practices as part of several clinical studies.26,31,34-37 Parents are using products to help care for their baby's skin and there is a need to help parents identify the most appropriate products through research. This study aims to help address this need.

ELIGIBILITY:
Inclusion Criteria:

Newborn babies:

* Healthy, full-term, male or female newborns (37+ weeks gestation), with healthy normal skin
* Newborn must be within 0-14 days old at Baseline for Phase 1 and within 0-28 days old at Baseline for Phase 2

Mothers:

* Mothers carrying singleton pregnancy of greater than or equal to (>=) 37-weeks gestation
* Mother is the one who regularly cares for the newborn. The mother must be available to attend every study visit
* Mother must be willing and able to participate in and comply with a study that requires using test products as directed on her newborn throughout study period
* Mother must be 18 years of age or older

Exclusion Criteria:

For both Newborn babies and Mother:

* History of a confirmed coronavirus disease 2019 (COVID-19) infection in the last 30 days
* Temperature >=38.0 degree Celsius (°C) /100.4-degree Fahrenheit (°F), measured
* Use of fever reducers within the past 2 days of each onsite visit. Exception: The use of fever reducers will be acceptable in this timeframe as long as it for the appropriate indication (example teething, immunization, etc.) and not COVID related as per principal investigator (PI) assessment
* Is participating in another clinical study where the participant is currently part of an active intervention/treatment (current or planned during the study period)

Newborn babies:

* Newborn has a chromosomal abnormality or other syndromic diagnosis
* Newborn has major congenital malformations or limb defects
* Newborn is currently admitted to a neonatal unit
* Newborn with health concerns
* Newborn with known allergies or adverse reactions to common topical skincare products
* Any condition requiring use of a topical or oral over the counter (OTC) or prescription medication, which in the investigator's judgment makes the subject ineligible or places the subject at risk. Child vitamins are allowed and should be listed on the Medical Information sheet (Health and Eligibility Questionnaire) under the Concurrent Medications section
* Newborn with a known condition of asthma or any related breathing problems
* Newborn with chronic medical conditions or treatments that could interfere with the study or pose a risk to the newborn (including known immunodeficiency or lung related conditions)
* Newborn with active localized or general infections including upper respiratory infections (ear, nose, throat, fever, cough, Et cetera [etc.]).
* Have been in close contact (exposure within 6 feet/2 meters for a cumulative 15 minutes or more over a 24-hr period) with anyone who has been infected with COVID-19 within the last 14 days or the newborn is under an isolation/quarantine order (prior to enrollment and visit 6)
* Per Mother's report of her newborn's symptoms within the past 2 weeks: Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness

Mother:

* Mother has a known allergies or adverse reactions to the ingredients of any of the test products
* Mother is unable to satisfactorily give informed consent for participation
* A social issue or logistical reason that, at the discretion of the direct care team, will prevent comfortable study participation by the family
* Have been in close contact (exposure within 6 feet/2 meters for a cumulative 15 minutes or more over a 24-hr period) with anyone who has been infected with COVID-19 within the last 14 days or is under an isolation/quarantine order (prior to enrollment and visit 6)
* Participants with self-reported symptoms within the past 2 weeks: Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Change in neonatal skin condition score from baseline to 3 weeks | 3 weeks
  Phase 1
Change in Transepidermal Water Loss (TEWL) from baseline to 12 weeks | 12 weeks
  Phase 2
Change in stratum corneum hydration (corneometer) from baseline to 12 weeks | 12 weeks
  Phase 2
Number of adverse events reported related to investigations products | 3 weeks
  Phase 1

SECONDARY OUTCOMES:
Product Questionnaires | 3 weeks
  Phase 1
Change in neonatal skin condition score from baseline to 12 weeks | 12 weeks
  Phase 2
Change in stratum corneum surface water content (ATR-FTIR) from baseline to 12 weeks | 12 weeks
  Phase 2
Change in stratum corneum lipid structure (ATR-FTIR) from baseline to 12 weeks | 12 weeks
  Phase 2
Change in stratum corneum carboxylate levels (ATR-FTIR, marker of natural moisturizing factor levels and filaggrin expression) from baseline to 12 weeks | 12 weeks
  Phase 2

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Saint Mary's Hospital, Manchester, Machester
  - The Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- See also: A Randomized Controlled Trial of Gentle Touch/Early Massage with a New Wash and Lotion Regimen for Improved Skin Barrier Strength, Parental Bonding, and Physical Development in Newborn Babies — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-1610%201411%202628-SBCT&attachmentIdentifier=3eb3cd03-868c-496a-b4d2-3e682f21823e&fileName=CO-161014112628-SBCT_CSR.pdf&versionIdentifier=